CLINICAL TRIAL: NCT03746951
Title: Comparative Evaluation of Lumbar Plexus and Suprainguinal Fascia Iliaca Compartment Blocks for Pain Management After Orthopedic Surgical Procedures Involving Hip and Femur in Pediatrics.
Brief Title: Comparative Evaluation of Lumbar Plexus and Suprainguinal Fascia Iliaca Compartment Blocks
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Senthil G. Krishna, Attending Anesthesiologist, Nationwide Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB18-01102
Record Dates: First submitted 2018-11-16; First posted 2018-11-20 (Actual); Results first posted 2022-03-03 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: Orthopedic Disorder
MeSH Terms: conditions — Musculoskeletal Diseases | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fascia iliaca compartment block (FICB) (Active Comparator): FICB is a local anesthetic nerve block, a type of local anesthesia, used for the hip, thigh, and knee. It is performed by inserting the needle into the groin.
  Interventions: Drug: Ropivacaine Hcl 0.5% Inj Vil 20Ml
- Lumbar plexus block (LPB) (Active Comparator): LPB is a local anesthetic nerve block, a type of local anesthesia, used for the hip, thigh, and knee. It is performed by inserting the needle into the back.
  Interventions: Drug: Ropivacaine Hcl 0.5% Inj Vil 20Ml

INTERVENTIONS:
Drug: Ropivacaine Hcl 0.5% Inj Vil 20Ml — Anesthetic agent used in peripheral nerve block
  Other Names: Naropin

SUMMARY:
The investigators aim to compare the use of a suprainguinal fascia iliaca compartment block vs lumbar plexus block as an adjunct to general anesthesia in pediatric patients undergoing orthopedic procedures involving the hip or upper femur. This study will help determine the efficacy of the two techniques and their advantages when compared to each other including time to perform the block, opioid consumption reduction, effects on postoperative pain, and the length of stay.

ELIGIBILITY:
Inclusion Criteria:

* ASA grade I-III
* Undergoing elective orthopedic surgical procedures involving the hip and upper thigh

Exclusion Criteria:

* Local anesthetic allergy
* Skin or localized infection at the site of catheter insertion
* Patient or parent refusal

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2019-04-24 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fascia Iliaca Compartment Block (FICB) | Lumbar Plexus Block (LPB)
Started | 8 | 7
Completed | 8 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fascia Iliaca Compartment Block (FICB) | Lumbar Plexus Block (LPB) | Total
Number analyzed (Participants) | 8 | 7 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8 | 7 | 15
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 14 [8 to 16] | 13 [7 to 16] | 13 [7 to 16]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 5 | 4 | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 8 | 7 | 15
Weight [Median (Inter-Quartile Range); unit: kilograms] | 63.7 [25.3 to 90.7] | 45 [23 to 67.5] | 59.7 [27 to 75]
Height [Median (Inter-Quartile Range); unit: centimeters] | 167.5 [118 to 179.7] | 150.4 [119.8 to 166.4] | 158 [122.7 to 177.1]

OUTCOME MEASURES:

1. Primary Outcome: Total Time to Perform the Regional Anesthesia Technique
Description: The amount of time if takes to perform either the FICB or LPB.
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Fascia Iliaca Compartment Block (FICB) | Lumbar Plexus Block (LPB)
Number analyzed (Participants) | 8 | 7
minutes | 3 [3 to 6] | 6 [4 to 11]

2. Secondary Outcome: Opioid Consumption in the PACU
Description: Total number of subjects that required opioids to control pain in the post-anesthesia care unit (PACU).
Time Frame: Immediately to 1 hour post-op
Measure: Number; unit: participants
Arm/Group | Fascia Iliaca Compartment Block (FICB) | Lumbar Plexus Block (LPB)
Number analyzed (Participants) | 8 | 7
participants | 7 | 5

3. Secondary Outcome: Post-op Pain Scores
Description: Pain scores during the post-operative recovery period. Pain score scale is 0-10 with 0 being no pain and 10 being worst pain imaginable.
Time Frame: 48 hours post-op
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Fascia Iliaca Compartment Block (FICB) | Lumbar Plexus Block (LPB)
Number analyzed (Participants) | 8 | 7
units on a scale | 2.95 [0 to 8] | 3.78 [0 to 10]

ADVERSE EVENTS:
Time Frame: 48 hours post-op
Arm/Group | Fascia Iliaca Compartment Block (FICB) | Lumbar Plexus Block (LPB)
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/7
Other Adverse Events (participants affected / at risk) | 0/8 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-06): https://cdn.clinicaltrials.gov/large-docs/51/NCT03746951/Prot_SAP_000.pdf